CLINICAL TRIAL: NCT01836614
Title: Intravenous Lidocaine Infusion in the Management of Post-operative Pain in Colorectal Patients
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study was closed due to recommendations of performing a PK study first.
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CCHMC 2012-0674
Record Dates: First submitted 2013-04-08; First posted 2013-04-22 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Colorectal Disorders
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lidocaine (Active Comparator): The treatment group will receive a 1.5mg/kg intravenous lidocaine bolus over 10 minutes. The bolus will be followed by an intravenous lidocaine infusion of 1 mg/kg/hr. The infusion will be stopped after extubation prior to leaving the operating room or after 5 hours from the start of the infusion
  Interventions: Drug: Lidocaine
- Saline (Placebo Comparator): The saline will be administered over an infusion pump over 10 minutes and followed by a bolus. The infusion will be stopped after extubation prior to leaving the operating room or after 5 hours from the start of the infusion.
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Lidocaine — The treatment group will receive a 1.5mg/kg intravenous lidocaine bolus over 10 minutes after induction by means of an infusion pump. This bolus will be followed by an intravenous lidocaine infusion of 1 mg/kg/hr. The infusion will be stopped after extubation prior to leaving the operative room or after 5 hours from the start of the infusion, which ever comes first.

SUMMARY:
The purpose of this study is to determine if an intravenous lidocaine infusion (compared to placebo) intraoperatively will decrease time to return of bowel function postoperatively, decrease postoperative pain, diminish postoperative opioid requirement, minimize inflammatory markers and shorten time to discharge after colorectal surgery.

DETAILED DESCRIPTION:
Lidocaine is an amide local anesthetic that has analgesic and anti-inflammatory properties. Lidocaine infusion is a very useful pain medication that is underutilized to treat surgical, chronic, and cancer pain in children. The investigators propose to examine the perioperative use of lidocaine infusion in children undergoing colorectal surgery that involves an abdominal incision. The investigators plan to measure the following outcomes: length of stay in hospital following abdominal surgery, postoperative pain scores, cumulative morphine consumption, incidences of opioid adverse-effects: respiratory depression, sedation, nausea, vomiting, time to passage of flatus, time to first bowel movement and end-tidal Sevoflurane in operating room throughout surgery. The following laboratory values will be measured: serial lidocaine levels of pharmacokinetics and safety levels, Pro- and anti-inflammatory cytokine measurements: IL-6, IL-8, IL-10, IL-1RA and genetic variants.

ELIGIBILITY:
Inclusion Criteria:

* male or female children 1-15 years of age
* ASA physical status 1-3
* scheduled for colorectal surgery with abdominal incision
* scheduled for complex urology surgical case

Exclusion Criteria:

* ASA physical status > 3
* postoperative intubation planned ahead of surgery
* history of chronic use of opioid
* history of hepatic,renal, or cardiac failure
* history of organ transplant
* BMI > 30
* history of cardiac arrhythmia
* history of long QT syndrome
* history of allergic reaction to lidocaine or similar agents
* history of seizure disorder
* patient without Peripherally Inserted Central Catheter or other central access with contraindication to inhalation induction
* family history or know patient susceptibility to malignant hyperthermia

Ages: 1 Year to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2015-01; Primary Completion 2018-03 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Length of stay in hospital following abdominal surgery | participants will be followed for the duration of hospital stay, an average of 1 week
  The primary outcome measure will be to monitor the length of stay in hospital following abdominal surgery.

SECONDARY OUTCOMES:
Postoperative pain scores | participants will be followed post-op, average 5 days
  Study staff will monitor patients pain every 15 minutes in the PACU and record documentation every 4 hours while on the floor.
Cumulative morphine consumption | participants will be followed post-op, average 5 days
  Staff will document how much morphine a patient uses post-operatively after abdominal surgery.
Incidences of opioid adverse-effects | participants will be followed post-op, average 5 days
  Study staff will monitor nursing notes for respiratory depression, sedation, nausea and vomiting
Time to passage of flatus and bowel movement | participants will be followed post-op, average 5 days
  Study staff will review nursing notes for time of passage of flatus and first bowel movement.
End-tidal Sevoflurane in operating room throughout surgery | participants will be measured until the end of the OR case, on average 6 hours
Serial lidocaine levels for pharmacokinetics and safety levels | participants will be measured until the end of the OR case, on average 6 hours and 24 hours post-operatively
  2 samples will be drawn at time of baseline IV placement Blood draw 0-3 minutes after bolus is complete Blood draw 9-15 minutes after the bolus is complete 2 blood samples will be drawn at the end of continuous infusion (either at end of surgery after extubation prior to leaving OR or after 5 hours from the start of the infusion) Blood draw 1 hour following the infusion Blood draw 2-3 hours following the end of the infusion 2 blood samples will be drawn 24 hours after surgery dependent of necessary labs
Pro- and anti-inflammatory cytokine measurements: IL-6, IL-8, IL-10, IL-1RA | participants will be measured until the end of the OR case, on average 6 hours and 24 hours post-operatively
  2 samples will be drawn at time of baseline IV placement Blood draw 0-3 minutes after bolus is complete Blood draw 9-15 minutes after the bolus is complete 2 blood samples will be drawn at the end of continuous infusion (either at end of surgery after extubation prior to leaving OR or after 5 hours from the start of the infusion) Blood draw 1 hour following the infusion Blood draw 2-3 hours following the end of the infusion 2 blood samples will be drawn 24 hours after surgery dependent of necessary labs
Genetic variants | participants will be measured until the end of the OR case, on average 6 hours and 24 hours post-operatively
  2 samples will be drawn at time of baseline IV placement Blood draw 0-3 minutes after bolus is complete Blood draw 9-15 minutes after the bolus is complete 2 blood samples will be drawn at the end of continuous infusion (either at end of surgery after extubation prior to leaving OR or after 5 hours from the start of the infusion) Blood draw 1 hour following the infusion Blood draw 2-3 hours following the end of the infusion 2 blood samples will be drawn 24 hours after surgery dependent of necessary labs

CONTACTS AND LOCATIONS:
Overall Officials: Smokey J Clay, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Background] Kaba A, Laurent SR, Detroz BJ, Sessler DI, Durieux ME, Lamy ML, Joris JL. Intravenous lidocaine infusion facilitates acute rehabilitation after laparoscopic colectomy. Anesthesiology. 2007 Jan;106(1):11-8; discussion 5-6. doi: 10.1097/00000542-200701000-00007. PMID 17197840
- [Background] Groudine SB, Fisher HA, Kaufman RP Jr, Patel MK, Wilkins LJ, Mehta SA, Lumb PD. Intravenous lidocaine speeds the return of bowel function, decreases postoperative pain, and shortens hospital stay in patients undergoing radical retropubic prostatectomy. Anesth Analg. 1998 Feb;86(2):235-9. doi: 10.1097/00000539-199802000-00003. PMID 9459225
- [Background] Candiotti KA, Yang Z, Morris R, Yang J, Crescimone NA, Sanchez GC, Bird V, Leveillee R, Rodriguez Y, Liu H, Zhang YD, Bethea JR, Gitlin MC. Polymorphism in the interleukin-1 receptor antagonist gene is associated with serum interleukin-1 receptor antagonist concentrations and postoperative opioid consumption. Anesthesiology. 2011 May;114(5):1162-8. doi: 10.1097/ALN.0b013e318216e9cb. PMID 21455057
- [Background] Yardeni IZ, Beilin B, Mayburd E, Levinson Y, Bessler H. The effect of perioperative intravenous lidocaine on postoperative pain and immune function. Anesth Analg. 2009 Nov;109(5):1464-9. doi: 10.1213/ANE.0b013e3181bab1bd. PMID 19843784
- [Background] Kuo CP, Jao SW, Chen KM, Wong CS, Yeh CC, Sheen MJ, Wu CT. Comparison of the effects of thoracic epidural analgesia and i.v. infusion with lidocaine on cytokine response, postoperative pain and bowel function in patients undergoing colonic surgery. Br J Anaesth. 2006 Nov;97(5):640-6. doi: 10.1093/bja/ael217. Epub 2006 Sep 4. PMID 16952918
- [Background] Harvey KP, Adair JD, Isho M, Robinson R. Can intravenous lidocaine decrease postsurgical ileus and shorten hospital stay in elective bowel surgery? A pilot study and literature review. Am J Surg. 2009 Aug;198(2):231-6. doi: 10.1016/j.amjsurg.2008.10.015. Epub 2009 Mar 12. PMID 19285304
- [Background] Bulloch B, Tenenbein M. Validation of 2 pain scales for use in the pediatric emergency department. Pediatrics. 2002 Sep;110(3):e33. doi: 10.1542/peds.110.3.e33. PMID 12205283
- [Background] McGrath PA, Seifert CE, Speechley KN, Booth JC, Stitt L, Gibson MC. A new analogue scale for assessing children's pain: an initial validation study. Pain. 1996 Mar;64(3):435-443. doi: 10.1016/0304-3959(95)00171-9. PMID 8783307
- [Background] Duedahl TH, Hansen EH. A qualitative systematic review of morphine treatment in children with postoperative pain. Paediatr Anaesth. 2007 Aug;17(8):756-74. doi: 10.1111/j.1460-9592.2007.02213.x. PMID 17596221
- [Background] Kain ZN, Mayes LC, Caldwell-Andrews AA, Karas DE, McClain BC. Preoperative anxiety, postoperative pain, and behavioral recovery in young children undergoing surgery. Pediatrics. 2006 Aug;118(2):651-8. doi: 10.1542/peds.2005-2920. PMID 16882820
- [Background] Annabi EH, Barker SJ. Severe methemoglobinemia detected by pulse oximetry. Anesth Analg. 2009 Mar;108(3):898-9. doi: 10.1213/ane.0b013e318172af73. PMID 19224799
- [Background] Ash-Bernal R, Wise R, Wright SM. Acquired methemoglobinemia: a retrospective series of 138 cases at 2 teaching hospitals. Medicine (Baltimore). 2004 Sep;83(5):265-273. doi: 10.1097/01.md.0000141096.00377.3f. PMID 15342970
- [Background] LUND PC, CWIK JC. PROPITOCAINE (CITANEST) AND METHEMOGLOBINEMIA. Anesthesiology. 1965 Jul-Aug;26:569-71. doi: 10.1097/00000542-196507000-00020. No abstract available. PMID 14313465